CLINICAL TRIAL: NCT07125924
Title: Intravesical Hyaluronic Acid (HA) for Preventing Radiation Cystitis on Bladder Cancer : A Randomized Controlled Trial
Brief Title: Intravesical Hyaluronic Acid (HA) for Preventing Radiation Cystitis on Bladder Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sung Uk Lee, M.D., Ph.D., National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: National Cancer Center, Korea
Record Dates: First submitted 2025-08-03; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer; Radiation Cystitis
Keywords: Hyaluronic acid; Radiation Cystitis; Intravesical treatment; Prevention
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Blad-Care (sodium hyaluronate 1.6%, 800 mg/50 mL, BioPlus Co., Ltd.)
  Interventions: Device: Blad-Care (sodium hyaluronate 1.6%, 800 mg/50 mL, BioPlus Co., Ltd.)
- Control group (Sham Comparator): Normal saline (N.S.)
  Interventions: Other: Normal Saline (NS)

INTERVENTIONS:
Device: Blad-Care (sodium hyaluronate 1.6%, 800 mg/50 mL, BioPlus Co., Ltd.) — Bladder instillation of Blad-Care (sodium hyaluronate 1.6%, 800 mg/50 mL, BioPlus Co., Ltd.) will be administered aseptically once weekly for a total of five times following each session of radiotherapy.
  Arms: Intervention group
Other: Normal Saline (NS) — Normal saline will be instilled into the bladder following the same schedule as the intervention group, i.e., five times after each radiotherapy session.
  Arms: Control group

SUMMARY:
To evaluate the efficacy and safety of intravesical hyaluronic acid (HA) instillation therapy for the prevention of radiation-induced cystitis in patients undergoing radiotherapy for bladder cancer.

DETAILED DESCRIPTION:
Study Design: Single-blind, Randomized, Controlled trial.

* Primary endpoint

  - To assess patient-reported outcomes (PROs) related to symptoms of radiation-induced cystitis in patients with bladder cancer undergoing radiotherapy.
* Secondary endpoint

  * To evaluate tumor control rates in patients with bladder cancer undergoing radiotherapy.
  * To assess the incidence and severity of radiation-induced cystitis using RTOG/EORTC criteria, CTCAE grading, and cystoscopic findings.
  * To compare healthcare costs between the treatment group receiving intravesical hyaluronic acid instillation and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic confirmed Muscle-Invasive Urothelial Carcinoma I. Clinical stage: T2-T4a MIBC II. No or limited nodal involvement (N0 or partial N1, only isolated or regional) III. No distant metastasis (M0) IV. Transurethral resection of bladder tumor (TURBT): Maximal TURBT is available > Most tumors must be resected, and residual disease should be minimized.

   V. Preserved bladder function is required: patients must have normal bladder capacity and maintain adequate voiding function.

   VI. Unifocal or localized tumor (except multifocal) VII. No extensive carcinoma in situ (CIS)
2. Age ≥ 19
3. Karnofsky performance score (KPS) ≥ 70 or ECOG performance status 0~2
4. Patients who are candidates for bladder-preserving therapy, specifically those scheduled to undergo concurrent chemoradiotherapy (CCRT) instead of radical cystectomy.
5. Patients scheduled to receive radiotherapy in combination with one or more of the following chemotherapeutic agents prior to study enrollment: Cisplatin-based chemotherapy (e.g. weekly cisplatin), Gemcitabine or 5-FU/mitomycin, in accordance with standard clinical practice.
6. Written informed consent obtained from the patients prior to study participation

Exclusion Criteria:

1. Present of distant metastasis (M1)
2. Tumor invasion beyond the bladder wall into adjacent organs (T4b)
3. Non-urothelial carcinoma (including histologic variant) or predominant of non-urothelial components in mixed histology
4. Medically inoperable status or poor general condition (ECOG performance status > 2)
5. History of active cystitis or recurrent urinary tract infections within the past 6 months
6. Known hypersensitivity to hyaluronic acid or related compounds
7. Any condition in which, in the investigator's judgment, administration of the study drug or procedure is deemed inappropriate
8. Pregnant or breastfeeding women, or women of childbearing potential who are unable or unwilling to use adequate contraception during the study period

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-08-22 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 12 months
  To assess patient-reported outcomes (PROs) related to symptoms of radiation-induced cystitis using the EORTC QLQ-BLM30 questionnaire (Korean version) in patients with bladder cancer undergoing radiotherapy.

SECONDARY OUTCOMES:
Tumor Control | 12 months
  To evaluate tumor control rates in patients with bladder cancer undergoing radiotherapy.
Radiation-induced cystitis | 12 months
  To assess the incidence and severity of radiation-induced cystitis using RTOG/EORTC criteria.
healthcare costs | 12 months
  To compare healthcare costs between the treatment group receiving intravesical hyaluronic acid instillation and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Uk Lee, MD, PhD, Principal Investigator — Center for Proton Therapy, National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No